CLINICAL TRIAL: NCT00277251
Title: Double-Blinded Controlled Trial of Alendronate for the Treatment of Childhood and Adolescent Glucocorticoid- Associated Osteopenia and Osteoporosis
Brief Title: Alendronate Osteoporosis Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Glaser Pediatric Research Network (Network); Elizabeth Glaser Pediatric AIDS Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 04-12-187R
Record Dates: First submitted 2005-07-07; First posted 2006-01-16 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Glucocorticoid-Associated Osteopenia and Osteoporosis
Keywords: Crohn's disease; systemic-onset juvenile rheumatoid arthritis; juvenile dermatomyositis; systemic lupus erythematosus (SLE); Mixed connective tissue disease (MCTD); vasculitis
MeSH Terms: conditions — Osteoporosis; Crohn Disease; Arthritis, Juvenile; Dermatomyositis; Lupus Erythematosus, Systemic; Mixed Connective Tissue Disease; Vasculitis | interventions — Alendronate

INTERVENTIONS:
Drug: Alendronate

SUMMARY:
This trial will test the hypothesis that among 20 children and adolescents from Children's Hospital, Boston with Crohn's disease, ulcerative colitis, systemic-onset juvenile rheumatoid arthritis, juvenile dermatomyositis, systemic lupus erythematosus, mixed connective tissue disease and vasculitis, treatment of glucocorticoid-associated osteopenia and osteoporosis with 18 months of alendronate (FOSAMAX®, Merck & Co., Inc.) will result in greater improvement in the mean change of individual AP spine bone mineral density (BMD) (gm/cm2) determined by dual energy X-ray absorptiometry (DXA) than treatment with 18 months of standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be diagnosed with either ulcerative colitis, Crohn's disease, systemic-onset juvenile rheumatoid arthritis, juvenile dermatomyositis, systemic lupus erythematosus (SLE), mixed connective tissue disease (MCTD) or vasculitis according to standard criteria where available, and according to treating physicians when not available.
* Subjects must have diminished AP lumbar spine (L1-L4) BMD by DXA (Hologic 4500) with a Z score ≤ -1.5 SD assessed within 8 weeks of the Baseline Visit.
* Subjects must have received daily, alternate day or weekly systemic glucocorticoid therapy for a minimum of six months total in their life-time.
* Subjects must be between the ages of 8 and 21 years, 11 months, at randomization. Although subjects younger than 8 years of age may be affected by osteoporosis, limited normative data prevents assignment of a BMD Z score for this group.
* Regarding subjects with child-bearing potential Females who have had at least one menstrual cycle must either be abstinent or must be using an effective method of birth control.

Exclusion Criteria:

* Current or recent (within 6 months) treatment with therapeutic doses of a bisphosphonate, calcitonin, human growth hormone, and heparin, all agents known to alter bone density
* A history of recent (within one year of screening) major upper gastrointestinal (GI) disease (above the jejunum), including, but not limited to, peptic ulcer, esophageal disease or active GI bleeding, or ever had surgery of the upper GI tract other than pyloroplasty. A history of abnormalities of the esophagus which delay esophageal emptying, such as stricture or achalasia
* Hyperthyroidism (suppressed thyroid stimulating hormone (TSH) and elevated free thyroxine (T4)), hyperparathyroidism (elevated parathyroid hormone (PTH)), malignancy, rickets, or osteomalacia (by history), all assessed within 8 weeks of the Baseline Visit.
* 25 (OH) vitamin D below 20 mg/L
* Planned or current pregnancy and/or breastfeeding
* Renal dysfunction defined as dependence on dialysis or a creatinine clearance < 35 ml/min, assessed within 4 weeks of the Baseline Visit. Creatinine clearance = [(height in cm x 0.55)/plasma creatinine] for all females and for males < 13 years old; [(height in cm x 0.70)/plasma creatinine] for males ³ 13 years old.
* Hepatic insufficiency defined as SGPT or SGOT greater than twice normal for age, assessed within 4 weeks of the Baseline Visit.
* Uncorrected hypocalcemia (ionized calcium>10% below age-adjusted range), assessed within 4 weeks of the Baseline Visit
* Known or suspected hypersensitivity to bisphosphonates
* Inability to follow instructions for dosing, including being unable to swallow the study medication with plain water first thing in the morning, stand or sit upright without any other food or beverage for at least 30 minutes following dosing and until their next meal
* Weight greater than 136 kg (300 lb), as the DXA is not reliable for subjects of this size
* Weight less than 17 kg (37 lb), assessed within 8 weeks of the Baseline Visit
* Permanent foreign body (prosthetic, surgical clips, permanent earring/umbilical ring) in region of results of the study
* Enrollment Procedures interest, or soft tissue calcinosis overlying the region of interest
* Inability to undergo dual energy X-ray absorptiometry or CT scan
* Developmental or cognitive delay which may interfere with cooperation and/or compliance with the procedures
* Subject expects to move out of the area during the study period, rendering follow-up per protocol impractical

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2003-03 (Actual); Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that among children and adolescents with Crohn's disease, ulcerative colitis, systemic-onset juvenile rheumatoid arthritis, juvenile dermatomyositis, systemic lupus erythematosus, mixed connective tissue disease and vasculitis, tr

SECONDARY OUTCOMES:
Alternate outcome measures
Comparison of DXA and QCT
Predictors for response to alendronate
Growth velocity
Fracture assessment

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Gordon, MD, Principal Investigator — Boston Children's Hospital